CLINICAL TRIAL: NCT01168947
Title: Effect of Sodium Concentration of Priming and Rinsing Fluids on Interdialytic Weight Gain and Blood Pressure in Hemodialysis Patients: a Prospective Pilot Study
Brief Title: Effect of Sodium Concentration of Priming and Rinsing Fluids on Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 052-10
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Fluid Overload and Hypertension in Hemodialysis Patients
Keywords: sodium; hypertension; fluid overload; hemodialysis; dialysate; interdialytic weight gain; intradialytic hypotension
MeSH Terms: conditions — Edema; Hypertension

ARMS (1):
- 5% dextrose (Experimental): 5% dextrose rinsing fluid
  Interventions: Other: 5% dextrose solution

INTERVENTIONS:
Other: 5% dextrose solution — The extracorporeal circuit of the dialysis machine will be primed and rinsed with a 5% dextrose solution instead of 0.9% saline.

SUMMARY:
Sodium loading during hemodialysis treatment is common and may contribute to increased interdialytic weight gain and hypertension. Excessive use of isotonic saline (containing 0.9% sodium chloride) is one of the factors that may cause sodium loading. During each hemodialysis session, approximately 400 mL of isotonic saline fluid, representing 1.4 grams of sodium, is used to prime and rinse the extracorporeal circuit, and is often administered to the patient. Switching to a non sodium-containing priming and rinsing fluid could allow for removal of the equivalent amount of sodium.

Switching to a non sodium-containing solution for the priming and rinsing of the extracorporeal circuit can contribute to increased sodium removal during the dialysis treatment and allow for reduced interdialytic weight gain, reduced thirst, and improved blood pressure control.

DETAILED DESCRIPTION:
This 12 week study consists of 3 phases:

Phase 1 (4 weeks): Observation only. Standard priming/rinsing procedure with isotonic saline Phase 2 (4 weeks): Intervention. Switch to a 5% dextrose solution for priming/rinsing procedure Phase 3 (4 weeks): Switch back to standard priming/rinsing procedure with isotonic saline During the study, blood pressures will be measured in a standardized manner at 2 week intervals, a thirst questionnaire will be completed at the end of each phase, and interdialytic weight gain, in-center pre/post-HD blood pressure and intradialytic symptoms will be recorded, apart for routinely measured parameters.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, clinically stable maintenance HD patients on a thrice weekly HD regimen.
* Willing and able to provide written, signed informed consent after the nature of the study has been explained.
* Willing and able to comply with all study procedures.
* Age ≥18 years.

Exclusion Criteria:

* Diabetes mellitus
* Considerable residual renal function (diuresis > 500 mL/day)
* Simultaneous participation in another clinical study except observational trials
* Any psychological condition which could interfere with the patient's ability to comply with the study protocol
* Expectation that native kidney function will recover
* Impossibility to perform a blood pressure measurement on the upper limb
* Unable to verbally communicate in English
* Scheduled for living donor kidney transplant, change to peritoneal dialysis, home HD or plans to relocate to another center during the study period.
* Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Interdialytic weight gain | 12 weeks

SECONDARY OUTCOMES:
Pre and post dialysis blood pressure levels. | 12 weeks
Intradialytic events. | 12 weeks
Thirst levels | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Yorkville Dialysis Center, New York, New York, United States

REFERENCES:
- [Derived] Rootjes PA, Penne EL, Ouellet G, Dou Y, Thijssen S, Kotanko P, Raimann JG. Dextrose solution for priming and rinsing the extracorporeal circuit in hemodialysis patients: A prospective pilot study. Int J Artif Organs. 2021 Nov;44(11):906-911. doi: 10.1177/03913988211020023. Epub 2021 May 31. PMID 34058888